CLINICAL TRIAL: NCT06411613
Title: Home-based Conservative Care Model for Advanced Kidney Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a budget deficit and hiring freeze, the intervention could not be implemented. Consequently, the study was modified from a pilot trial to an observational study.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 21-061
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases
Keywords: CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Test the feasibility and acceptability of a novel care program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CC Program Received Intervention (Experimental): The CC Program will be delivered through the existing HBPC infrastructure at VA Puget Sound Health Care System. Each HBPC team is comprised on a lead physician or nurse practitioner, nurse, pharmacist, nutritionist, social worker, psychologist, therapist, and chaplain. At a minimum, subsequent clinical encounters and assessments for each Veteran will be scheduled no less than on a quarterly basis and more often as needed based on the HBPC team's clinical judgment. On a monthly basis, the entire HBPC team will conduct MDC meetings to review each Veteran's medical plan. The Program aims to provide patient-centered, whole-person and team-based care, shared decision-making, active symptom management, advance care planning and end-of-life care.
  Interventions: Other: CC Program
- Usual Care (No Intervention): Does not receive intervention.

INTERVENTIONS:
Other: CC Program — The CC Program will be delivered through the existing HBPC infrastructure at VA Puget Sound Health Care System. Each HBPC team is comprised on a lead physician or nurse practitioner, nurse, pharmacist, nutritionist, social worker, psychologist, therapist, and chaplain. At a minimum, subsequent clinical encounters and assessments for each Veteran will be scheduled no less than on a quarterly basis and more often as needed based on the HBPC team's clinical judgment. On a monthly basis, the entire HBPC team will conduct MDC meetings to review each Veteran's medical plan. The Program aims to provide patient-centered, whole-person and team-based care, shared decision-making, active symptom management, advance care planning and end-of-life care.
  Arms: CC Program Received Intervention

SUMMARY:
This is a randomized pilot study to test the feasibility and acceptability of a novel conservative care (CC) pathway among patients with advanced chronic kidney disease (CKD) who have chosen to forgo initiation of maintenance dialysis, their caregivers and providers.

DETAILED DESCRIPTION:
This study is a randomized pilot study to test the acceptability and feasibility of a CC pathway, called the Kidney Care at Home Program, with patients with advanced CKD who have chosen to forgo dialysis, their caregivers and providers. The novel CC program will be developed upon an existing home-based multidisciplinary care (MDC) program in the Veterans Affairs (VA) called the Home-Based Primary Care (HBPC) program. HBPC provides for Veterans with multimorbidity and functional limitation with the goal of supporting Veterans' quality of life and mitigating the complications of illness through to the end of life.

The investigators hypothesize that HBPC serves as the ideal starting ground to build the VA's first CC program for Veterans with advanced CKD. The investigators will use implementation science and ethnographic research methods, including field observations, interviews, medical record review, and serial structured surveys on quality of life, symptom burden, care satisfaction and goal concordant care to assess the feasibility and acceptability of the Kidney Care at Home Program (intervention) vs. usual care (control).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Receives primary +/- nephrology care from VAPS as defined as having at least 1 outpatient primary or nephrology visit in the prior year
* Advanced CKD as defined as defined as having 2 or more outpatient measures of an eGFR 20 ml/min/1.73m2 separated by 90 or more days
* Unsure or do not wish to undergo maintenance dialysis
* Agreement by their VA primary +/- nephrology care provider that patients can participate in the study

Caregivers:

* Nominated by enrolled patient as a caregiver whom patient agrees to participate in the study

Clinicians:

* Employed at VAPS
* Identified by enrolled Veterans as important to their CKD and nominated by the Veteran to be interviewed for the study

Exclusion Criteria:

Patients:

* Unable to complete "teach-back" method of informed consent
* Currently receiving maintenance dialysis
* Currently enrolled in HBPC Program

Caregivers:

* Unable to complete "teach-back" method of informed consent
* If a Veteran withdraws from the study, their caregivers' participation in the study is also terminated at that time

Clinicians:

* If a Veteran withdraws from the study, their clinicians will no longer be eligible to participate in interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. O'Hare, MD MA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data collected and study protocols will be shared immediately following publication and ending 5 years following article publication with researchers who provide a written request and sound research proposal that has undergone human subjects review. Interested researchers can contact the principal investigator directly.
Supporting Information: Study Protocol
Time Frame: Available immediately following publication, ending 5 years following article publication.
Access Criteria: Available immediately following publication, ending 5 years following article publication.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only patients with advanced CKD were enrolled in the study. Caregivers and clinicians were not enrolled.
Period: Overall Study
Arm/Group | CC Program Received Intervention | Usual Care
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CC Program Received Intervention | Usual Care | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Interviews
Description: At each study visit, patients will be invited to complete a 45- to 60-minute interview to ascertain their experiences with and perspectives on their kidney care. Interviews will follow a structured guide intended to elicit: 1) benefits; 2) challenges; 3) unanticipated issues; and, 4) opportunities to improve respective approaches to care. Non-specific probes will be used to prompt subjects to elaborate on their responses for greater depth and detail. Veterans will be interviewed separately, in private, and in-person or by phone according to each person's preference. All interviews will be audio-recorded then transcribed without personal identifiers.
Time Frame: 1 year
Population: Due to a budget deficit and hiring freeze, the intervention could not be implemented and will not be collected in the future.
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Clinician Interviews
Description: Clinicians will be invited to participate in up to two 30-minute structured interviews about their perception of their experiences with and perspectives on patients' kidney care.
  Interviews will follow a structured guide similar to that for Veterans and caregivers.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Field Observations
Description: Patients will invite study staff to observe clinical encounters that they perceive as important to their kidney care.
  These clinical encounters can include face-to-face, telephone, and video encounters. During the encounter, study staff will either digitally audio-record and/or note-take conversations and interactions or only observe and note-take after the encounter per each subject's preference. After the encounter is complete, we will ask subjects clarifying questions about the encounter as needed
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Document Review
Description: Clinical progress notes entered into each patient's electronic medical record during the study period and abstract passages documenting care considerations regarding CKD.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Caregiver Interviews
Description: At each study visit caregivers of patients will be invited to complete a 45- to 60-minute interview to ascertain their experiences with and perspectives on the patient's kidney care.
  Interviews will follow a structured guide intended to elicit: 1) benefits; 2) challenges; 3) unanticipated issues; and, 4) opportunities to improve respective approaches to care. Non-specific probes will be used to prompt subjects to elaborate on their responses for greater depth and detail. Caregivers will be interviewed separately, in private, and in-person or by phone according to each person's preference. All interviews will be audio-recorded then transcribed without personal identifiers.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Health Outcomes Prioritization Scale
Description: At each study visit, patients will be asked to rank their health priorities and whether they receive care that is aligned with their top priority using the Health Outcomes Prioritization Scale: priority score 0-100 of four universal health outcomes: keeping you alive, maintaining independence, reducing or eliminating pain, and reducing or eliminating other symptoms, with higher scores indicating that the outcome was more important.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Zarit Burden Interview
Description: At each study visit, caregivers will be asked about caregiver strain: a 12 item survey asking caregivers to rate the frequency with which they experience different forms of caregiver strain using the Zarit Burden Interview (4-point scale which describes degree of burden experienced from 0=never to 4=almost always).
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Consultation Satisfaction Questionnaire
Description: At each study visit patients will be ask to rate their level of satisfaction with the care they receive using the Consultation Satisfaction Questionnaire. The Consultation Satisfaction Questionnaire is a 17-item survey utilizing Likert Scale responses: strongly disagree, somewhat disagree, neutral, somewhat agree, strongly agree, to assess overall care, professionalism, communication, time spent, and depth of the relationship with clinicians involved in their kidney care based on their last clinical visit.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Edmonton Symptom Assessment Scale
Description: At each study visit, patients will be asked about the presence and severity of common symptoms of advanced CKD using the Edmonton Symptom Assessment Scale (numeric rating scale 0=no symptoms to 10=worst possible).
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: EQ-5D-5L
Description: At each study visit, patients will be asked to rate different domains of their quality of life and overall health using the EuroQol 5D Questionnaire (EQ-5D-5L) to assess health-related quality of life. The EQ-5D-5L consists of two parts:
  1. EQ-5D Descriptive System: Includes Five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has five levels of severity ranging from no problems to extreme problems. The respondent indicates their health state by selecting the most appropriate level for each dimension.
  2. EQ Visual Analogue Scale (EQ-VAS): a scale where respondents rate their overall health from The worst health you can imagine (0) to the best health you can imagine (100).
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Non-Enrollment: Provider Did Not Agree to Recruitment of Veteran
Description: The investigators will record reasons why eligible Veterans' primary care +/- nephrology provider did not agree to recruitment of Veterans to participate in the study.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Non-Enrollment: Veteran Refusal to Participate
Description: The investigators will record reasons for refusal to participate in the study by eligible Veterans.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Attrition
Description: The investigators will ask enrolled subjects who withdraw from the study their reasons for withdrawal.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | CC Program Received Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline
Description: Discontinuity of care
Arm/Group | CC Program Received Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT06411613/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT06411613/ICF_000.pdf